CLINICAL TRIAL: NCT04487314
Title: Russian Registry for Chronic Venous Disease Incidence and Natural Course
Brief Title: Registry for Chronic Venous Disease Incidence and Natural Course
Acronym: RRCVD
Status: Recruiting | Type: Observational
Sponsor: Russian Phlebological Association (Other)
Responsible Party: Principal Investigator, Evgeny Ilyukhin, Principal Investigator, Russian Phlebological Association
Other Study IDs: RPA 10.001
Record Dates: First submitted 2020-07-09; First posted 2020-07-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Varicose Veins of Lower Limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without Chronic Venous Disease: Individuals who do not have signs of chronic venous diseases of lower legs according to Clinical, Etiologic, Anatomic and Pathophysiologic classification (CEAP)
- Patients with Chronic Veinous Disease: Individuals who have signs of chronic venous diseases of lower legs according to CEAP classification (telangiectases, varicose veins, venous edema, skin hyperpigmentation, lipodermatosclerosis, venous ulcer).

SUMMARY:
A prospective cohort study of patients with primary varicose veins to assess the morbidity, risk factors and development of chronic lower limb vein disease.

DETAILED DESCRIPTION:
Multicenter prospective cohort observational study based on a termless epidemiological registry.

Periodic inspection and collection of data from the subjects is carried out annually, in the last quarter of the current year.

Patient data is recorded in a promising digital database and is constantly updated.

ELIGIBILITY:
Inclusion Criteria:

* A family members of the researcher (spouse, childrens, brothers and sisters, parents) or the researcher himself
* The possibility of annual clinical and ultrasound assessment of the venous system of the observed individuals

Exclusion Criteria:

* Any invasive treatment of the chronic venous disorder in anamnesis
* Venous thrombosis in the anamnesis or at the time of inclusion

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The main cohort is formed from those who do not have CVD, who are affected by different factors that we register (various physical activities, the presence or absence of pregnancy, etc.).
  An additional cohort is formed from those who have CVD at the time of inclusion.
  The goal is to track the natural evolution (progression) of the disease, to evaluate the incidence and risk factors of complications.
  An extremely important criterion for the formation of the study population is the possibility to control the lower legs veins of observed individuals by a qualified vascular specialist. To date, a qualitative assessment of veins according to the CEAP classification is a weak point in longitudinal epidemiological studies.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2050-09-01 (Estimated); Study Completion 2050-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Chronic Venous Disease | 1 year
  Number of Participants with the first identified signs of chronic venous disease according to CEAP classification (telangiectasia, varicose veins, edema)
Natural Course of Chronic Venous Disease | 1 year
  Progression of CVD will be measured as a change in clinical class of CVD according to CEAP classification in every individual affected by CVD
Incidence of chronic venous insufficiency | 1 year
  Number of Participants with the first identified sign of chronic venous insufficiency (venous edema, venous eczema, hyperpigmentation of the skin, lipodermatosclerosis, venous ulcer)
Incidence of superficial vein thrombosis | 1 year
  Number of Participants with the first identified sign of superficial vein thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- "Medalp" private surgery clinic, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This is a website specially created for this register. — https://epid.venousregistry.org/
- See also: The Association of Phlebologists of Russia already has 2 registers, which registered in ClinicalTrials.gov and on the basis of which clinical trials are conducted. — https://www.venousregistry.org/